CLINICAL TRIAL: NCT07265817
Title: Fecal Microbiota Transplantation for Decolonization of Multidrug-resistant Microorganisms: Randomized Double Blinded Study
Brief Title: Fecal Microbiota Transplantation for Decolonization of Multidrug-resistant Microorganisms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Eun Soo Kim, MD, PhD, Professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KNUH 2023-07-013
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Carbapenem-Resistant Enterobacteriaceae Colonization

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal microbiota transplantation group (Active Comparator)
  Interventions: Combination Product: Fecal Microbial transplant Capsules
- Placebo (Placebo Comparator)
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: Fecal Microbial transplant Capsules — 3 pills per day for 3 consecutive days with placebo comparatator
  Arms: Fecal microbiota transplantation group
Combination Product: Placebo — The same amount and shape capsules
  Arms: Placebo

SUMMARY:
The aim of the study is to see whether fecal microbiota transplantation is effective to decolonize multidrug-resistant organisms.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have positive results in PCR or culture of rectal swab.

Exclusion Criteria:

* Not provide a consent.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Conversion to negative organism | 1 year

IPD SHARING:
Plan to Share IPD: No